CLINICAL TRIAL: NCT03052972
Title: Flortaucipir (18F) PET Imaging in the BIOCARD Study
Brief Title: Flortaucipir 18F PET Imaging in BIOCARD Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study terminated due to lower than expected enrollment
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A20
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amyloid Positive (Experimental): Clinically normal amyloid positive subjects from BIOCARD study receiving a flortaucipir PET scan
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Amyloid Negative (Experimental): Clinically normal amyloid negative subjects from BIOCARD study receiving a flortaucipir PET scan
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq)(10 millicurie [mCi]) single dose
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This study is designed to assess the imaging characteristics of Flortaucipir (18F-AV-1451) in subjects who participated in the Biomarkers of Cognitive Decline Among Normal Individuals (BIOCARD) study at Johns Hopkins University.

ELIGIBILITY:
Inclusion Criteria:

* Males or females that have provided consent and are currently enrolled in BIOCARD study
* Ability to tolerate PET scan procedures
* Ability to provide informed consent for study procedures

Exclusion Criteria:

* Has condition(s) that could augment risk to participant or compromise ability to tolerate experimental procedures or interfere with analysis of the study data as determined by the investigator
* Has a history of risk factors for Torsades de Pointes or taking medications known to cause QT prolongation.
* Has electrocardiogram acquired prior to initial flortaucipir scan that clinically contradicts subject's participation in the study as determined by the investigator. Bazett's corrected QT (QTcB) interval must be assessed and not exceed accepted values (458 msec in males, 474 msec in females).
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity, or not using reliable contraceptive methods.
* Has hypersensitivity to flortaucipir
* Has a currently clinically significant infectious disease, endocrine/metabolic disease, pulmonary/renal/hepatic impairment, or cancer that could impact study participation or scan results in the opinion of the investigator.
* Has a non-study related radiopharmaceutical imaging/treatment procedure within seven days prior to flortaucipir imaging visit.
* Is unsuitable for a study of this type in the opinion of the investigator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- See also: BIOCARD Study Summary — https://www.jhsph.edu/faculty/research/search/results/project/8899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place between Mar 2017 and Aug 2018 from the Biomarkers of Cognitive Decline Among Normal Individuals (BIOCARD) study
Period: Overall Study
Arm/Group | Amyloid Positive | Amyloid Negative
Started | 18 | 5
Completed | 18 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amyloid Positive: Clinically normal amyloid positive subjects from BIOCARD study
- Amyloid Negative: Clinically normal amyloid negative subjects from BIOCARD study
- Total: Total of all reporting groups
Arm/Group | Amyloid Positive | Amyloid Negative | Total
Number analyzed (Participants) | 18 | 5 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (5.69) | 66.8 (7.53) | 70.9 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 5 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 5 | 23
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 29.3 (1.02) | 29.2 (1.30) | 29.3 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Evaluation of Scan Results
Description: Subject scans were visually evaluated by an expert reader into three groups. Advanced Alzheimer's disease (AD) scan pattern = In either hemisphere, increased neocortical activity in the parietal/precuneus region(s), or frontal region(s) with increased uptake in the posterolateral temporal (PLT), parietal, or occipital region(s). Moderate AD scan pattern = In either hemisphere, increased neocortical activity limited to the PLT or occipital region(s). Not AD scan pattern = No increased neocortical activity, or increased neocortical activity isolated to the mesial temporal, anterolateral temporal, and/or frontal regions.
Time Frame: Baseline scan
Population: Subjects with visually evaluable PET scans (n=22). One scan was considered unevaluable by the expert reader.
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloid Positive | Amyloid Negative
Number analyzed (Participants) | 17 | 5
Participants
  Advanced AD Scan Pattern (τAD++) | 11 | 0
  Moderate AD Scan Pattern (τAD+) | 0 | 0
  Not AD Scan Pattern (τAD-) | 6 | 5

2. Primary Outcome: Quantitative Evaluation of Scan Results
Description: Standard Uptake Value Ratio (SUVr) by amyloid status using a weighted cortical average. For SUVr, a value of 1 or lower signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: 75 minutes post dose administration
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Groups:
- Total: All subjects from BIOCARD study receiving a flortaucipir PET scan
Arm/Group | Amyloid Positive | Amyloid Negative | Total
Number analyzed (Participants) | 18 | 5 | 23
standardized uptake value ratio (SUVr) | 1.0414 (0.04165) | 1.0219 (0.02057) | 1.0371 (0.03854)

ADVERSE EVENTS:
Time Frame: AEs were collected at scan visits and for 48 hours after flortaucipir administration.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection, at an imaging visit. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Arm/Group | Amyloid Positive | Amyloid Negative
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/5
Other Adverse Events (participants affected / at risk) | 2/18 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amyloid Positive (N=18) | Amyloid Negative (N=5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to slower than expected enrollment, the study was terminated before 100 subjects were recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03052972/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03052972/SAP_001.pdf